CLINICAL TRIAL: NCT00737776
Title: NovoMix® 30 UPGRADE (NovoMix® 30 Use for Progressed Glycemic Control in Realistic Administration to DiabEtes Mellitus): A Multicentre, Open Label, Nonrandomised, Non-interventional, Observational, Efficacy and Safety Study in Patients Using Biphasic Insulin Aspart 30 (NovoMix® 30) for the Treatment of Diabetes Mellitus
Brief Title: Observational Study on Efficacy and Safety in Patients Using NovoMix® 30 for the Treatment of Diabetes
Acronym: UPGRADE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3547
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoMix® 30; NovoLog® Mix 70/30

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the efficacy on blood glucose control while using NovoMix® 30 FlexPen® under normal clinical practice conditions in Korea. A clinical safety profile will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with type 1 and type 2 diabetes who are treated with NovoMix® 30
* Patient who signed on informed consent form

Exclusion Criteria:

* Patients who are unlikely to comply with protocol requirements, e.g., uncooperative attitude, inability to return for the final visit
* Patients who were previously enrolled in this study
* Patients with a hypersensitivity to NovoMix® 30 or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with type 1 and type 2 diabetes who are prescribed with NovoMix® 30
Sampling Method: Non-Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
HbA1c change | at the end of study after 26 weeks

SECONDARY OUTCOMES:
Number of serious adverse drug reactions | during the study
Number of serious adverse events | during the study
Number of all major (daytime and nocturnal) hypoglycaemic events | during the study
Number of major hypoglycaemic events related to omission of a meal after NovoMix® 30 injection | during the study
Number of major hypoglycaemic events related to physical exercise of at least 30 min | during the study
Number of all minor (daytime and nocturnal) hypoglycaemic events | during the study
Weight (BMI) change | at the end of study after 26 weeks
Lipid profile (Total cholesterol, LDL, HDL, Triglyceride) change | at the end of study after 26 weeks
Percentage of patients reaching the target of HbA1c below or equal to 6.5% | at the end of study after 26 weeks
Percentage of patients reaching the target of HbA1c below or equal to 7.0% | at the end of study after 26 weeks
Percentage of patients reaching the physician's own target recommendation | at the end of study after 26 weeks
Variability in fasting plasma glucose values and average (mean) fasting plasma glucose level | at the end of study after 26 weeks
Average post-breakfast (2h), post-lunch (2h), post-dinner (2h) plasma glucose level | at the end of study after 26 weeks
Diabetes Fear of Self-Injection Questionnaire (D-FISQ) | at the end of study after 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com